CLINICAL TRIAL: NCT04558112
Title: Improving Therapeutic Learning for PTSD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019-1567; SMPH/PSYCHIATRY/PSYCHIATRY (Other: UW Madison); 4R33MH108753-03 (NIH); A538900 (Other: UW Madison); Protocol Version 6/26/2023 (Other: UW Madison)
Record Dates: First submitted 2020-09-15; First posted 2020-09-22 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-07

CONDITIONS: PTSD; Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Levodopa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 100 mg L-DOPA (Experimental): Complete a ~40 min fMRI scan with either hearing their trauma or neutral narrative, ingest a pill (placebo or 100mg L-DOPA) upon leaving the scanner and wait in a waiting room for ~45 minutes, then undergo a 7 min resting-state fMRI scan.Participants return ~24 hours later for Day 2 fMRI, in which they will complete a single ~40-minute fMRI scan while listening to either their trauma or neutral narrative.
  Interventions: Drug: L-DOPA
- Placebo (Placebo Comparator): Complete a ~40 min fMRI scan with either hearing their trauma or neutral narrative, ingest a pill (placebo or 100mg L-DOPA) upon leaving the scanner and wait in a waiting room for ~45 minutes, then undergo a 7 min resting-state fMRI scan.Participants return ~24 hours later for Day 2 fMRI, in which they will complete a single ~40-minute fMRI scan while listening to either their trauma or neutral narrative.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: L-DOPA — two gel capsules with 100mg L-DOPA (with 25 mg carbidopa to inhibit peripheral decarboxylase)
  Arms: 100 mg L-DOPA
Drug: Placebo — two gel capsules of placebo
  Arms: Placebo

SUMMARY:
The proposed project seeks to demonstrate the engagement of post-exposure dopamine neurotransmission and downstream acute reorganization of dopaminergic resting-state neural networks as a means of increasing consolidation of extinction memories formed during analogue exposure therapy in adult women with PTSD. Participants will include 120 women aged 21-50 with a current diagnosis of PTSD related to physical or sexual assault, English speaking, and medically healthy. Participants will complete the stages of the study across 2-3 days, depending on participant need.

DETAILED DESCRIPTION:
Specific Aim 1: Test the degree to which exogeneous manipulations of dopamine neurotransmission affect exposure therapy learning across multiple indices. Hypothesis: L-DOPA will decrease measures of fear responding across indices.

Specific Aim 2: Test the degree to which post-exposure functional connectivity within dopaminergic neural networks mediates the effect of dopaminergic manipulation on fear responding after exposure therapy. Hypothesis: L-DOPA will predict enhanced post-exposure dopaminergic functional connectivity, which in turn predicts decrease fear recall.

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis of PTSD where the index traumatic event includes physical or sexual assault
* English speaking
* Medically healthy

Exclusion Criteria:

* internal ferromagnetic objects (such as electronic devices, surgical implants, shrapnel, etc.)
* major medical disorders (such as cancer)
* psychotic disorders
* neurocognitive disorders
* developmental disorders
* pregnancy
* breastfeeding
* use of Monoamine oxidase inhibitors (MAO-I) in past two weeks is exclusionary

Additional Exclusion Criteria at UT-Austin:

* heart disease
* hepatic impairment
* peptic ulcer disease
* COPD
* prescription medications that may interact with L-DOPA will not be permitted during a predetermined wash-out period

Due to safety concerns, participants with these conditions will be ineligible to participate:

* Claustrophobia, or the inability to lie still in a confined space
* Major medical disorders (e.g., HIV, cancer)
* Magnetic metallic implants (such as screws, pins, shrapnel remnants, aneurysm clips, artificial heart valves, inner ear (cochlear) implants, artificial joints, and vascular stents), as these may heat, pull, or twist in the strong magnetic field of the MRI scanner
* Electronic or magnetic implants, such as pacemakers, as these may stop working
* Permanent makeup or tattoos with metallic dyes
* A positive pregnancy test (for females), since the effect of strong magnetic fields and L-Dopa on the developing fetus remains unknown and inconclusive. (all female participants of childbearing potential will have a pregnancy test on the day of the MRI scan. Participants who test positive would be notified of this positive result)
* A self-reported history of loss of consciousness (greater than 30 minutes)
* Physical disabilities that prohibit task performance (such as blindness or deafness)
* Psychotic disorders (e.g., schizophrenia)
* Any other condition that the investigator believes might put the participant at risk

Due to their effects on image quality, participants with the following MAY be ineligible to participate per Principal Investigator's judgment:

* Medications which may affect image quality (e.g., water pills)
* Nonremovable dental implants, such as braces or upper permanent retainers, as these will distort the MRI images we collect (note: filings, crowns, and silver or gold teeth are OK)
* Any other condition, medication, or implant that the investigator believes would degrade image quality or render data unusable

Ages: 21 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2021-02-18 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change in negative emotional responding to trauma scripts on Day 2 compared to Day 1 | up to 2 days
  Measured periodically through the narrative with a 10-point Likert scale of anxiety/distress (self-reported), with higher numbers indicating increased anxiety/distress. Measured on day 1 and day 2

SECONDARY OUTCOMES:
Change in Skin Conductance Response (SCR) to trauma scripts on Day 2 compared to Day 1 | up to 2 days
  SCR data will be acquired on a BIOPAC MP150 Data Acquisition System (BIOPAC Systems, Inc.) with electrodes placed on participant's left hand. Average intensity of participant skin conductance will be reported. Measured on day 1 and day 2
Change in Heart Rate (HR) to trauma scripts on Day 2 compared to Day 1 | up to 2 days
  Heart rate data will be acquired with a pulse oximeter placed on participant's left hand. Average intensity of participant heart rate will be reported. Measured on day 1 and day 2
Change in amygdala-hippocampus functional connectivity on Day 2 compared to Day 1 | up to 2 days
  Measured by 3T functioning magnetic resident imaging (fMRI), time courses of activity of the hippocampus and amygdala will be correlated on day 1 and day 2, then compared between the groups.

CONTACTS AND LOCATIONS:
Overall Officials: Zachary Stowe, MD, Principal Investigator — University of Wisconsin, Madison
Locations (2):
- United States (2):
  - University of Texas, Austin, Texas
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No